CLINICAL TRIAL: NCT03836716
Title: Open Label, Non-randomized Extension Trial to Assess Long Term Safety and Efficacy of Arimoclomol in Subjects With Amyotropic Lateral Sclerosis Who Have Completed the ORARIALS-01 Trial
Brief Title: Arimoclomol in Amyotropic Lateral Sclerosis - Open Label Extension Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: As a consequence of the results of ORARIALS-01 which did not meet any of its efficacy endpoints. The planned duration was 152 weeks. After termination, the actual mean duration of treatment was approx. 28 weeks (range approx. 2 to 71 weeks).
Sponsor: ZevraDenmark (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORARIALS-02
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Arimoclomol; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — arimoclomol

STUDY DESIGN:
Intervention Model Description: Non-randomized open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arimoclomol (Experimental): 248 mg arimoclomol base (equivalent to 400 mg arimoclomol citrate) 3 times daily
  Interventions: Drug: Arimoclomol

INTERVENTIONS:
Drug: Arimoclomol — 2 capsules (2 x 124 mg arimoclomol base; equivalent to 2 x 200 mg arimoclomol citrate) taken 3 times daily

SUMMARY:
A multicenter, non-randomized, open label trial, to assess long term safety and efficacy of Arimoclomol in subjects with Amyotrophic Lateral Sclerosis (ALS) who have completed the ORARIALS-01 trial.

DETAILED DESCRIPTION:
The planned duration of the open-label trial was 152 weeks, but the trial was terminated early as a consequence of the results of ORARIALS-01 which did not meet any of its efficacy endpoints. Therefore, the actual mean duration of open-label treatment was approximately 28 weeks (range approximately 2 to 71 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to comprehend and is willing to provide written informed consent and is capable and willing to comply with trial procedures, or in the circumstance that the subject is incompetent, informed consent/assent is provided in accordance with local regulation and/or procedures
* Subject has completed the ORARIALS-01 trial (i.e., met one of the surrogate survival endpoints of tracheostomy or PAV or has completed the 76 weeks randomized treatment period)
* Subject completed ORARIALS-01 while on treatment, where on treatment is defined as having taken the last dose of IMP within 2 weeks of the End of Trial visit (whether at week 76 or prior)

Exclusion Criteria:

* Known or suspected allergy or intolerance to the IMP (Arimoclomol or constituents)
* Exposure to any other investigational treatment, advanced therapy medicinal product or use of any other prohibited concomitant medications
* Women who are lactating or pregnant, or men or women unwilling to use a highly effective method of birth control if not surgically sterile (defined as bilateral tubal ligation, bilateral oophorectomy, or hysterectomy for women; vasectomy for men) for female participants until 4 weeks after last dose and for male participants until 3 months after last dose. Pre-menopausal women must have a negative pregnancy test prior to dosing with trial medication.
* Any of the following medically significant conditions:

  1. Clinically significant renal or hepatic disease OR clinical laboratory assessment (results ≥ 3 times the upper limit of normal [ULN] for aspartate aminotransferase and/or alanine aminotransferase, bilirubin ≥ 2 times the ULN, or creatinine ≥ 1.5 times the ULN).
  2. Any new condition or worsening of existing condition which, in the opinion of the investigator, would put the subject at undue risk.
* Any serious adverse event or moderate/severe adverse event from the ORARIALS-01 trial which is ongoing at the time of transitioning to ORARIALS-02 and assessed as probably related to IMP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benatar, MD PhD, Principal Investigator — University of Miami
Locations (23):
- United States (7):
  - St. Joseph's Hospital and Medical Center (SJHMC) - Barrow Neurological Institute (BNI) - The Gregory W. Fulton ALS and Neuromuscular Disease Center, Phoenix, Arizona
  - UC Irvine Health ALS and Neuromuscular Center, Orange, California
  - University of Miami, Miami, Florida
  - Hospital for Special Surgery, New York, New York
  - Providence Brain & Spine Institute, Portland, Oregon
  - University of Pensylvania, Perelman Center for Advanced Medicine - Penn Neuroscience Center, Philadelphia, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
- Catholic University Leuven, Leuven, Belgium
- London Health Sciences Centre, London, Ontario, Canada
- France (2):
  - Centre Hospitalier Regional Universitaire (CHRU) Montpellier - Hopital Gui De Chauliac, Montpellier
  - Groupe Hospitalier Pitie-Salpetriere - Centre d'Investigation Clinique Neurosciences 1422, Paris
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum (CVK) - Ambulanz fuer ALS und andere Motoneuronenerkrankungen, Berlin
  - Medizinische Hochschule Hannover (MHH) - Klinik fuer Neurologie, Hanover
  - Universitaetsklinikum Ulm - Klinik fuer Neurologie, Ulm
- Italy (2):
  - Instituti Clinica Scientifici Maugeri, Milan
  - Azienda Ospedaliero Universitaria (AUO) di Torino - Citta'della Salute e della Scienza di Torino, Torino
- University Medical Center Utrecht, Utrecht, Netherlands
- Poland (2):
  - Centrum Medyczne NeuroProtect, Warsaw
  - Citi Clinic, Warsaw
- Spain (2):
  - Hospital Universitario Vall d'Hebron ALS Unit. Consultas Externas; Office: 9-10-11, Barcelona
  - Hospital Carlos III - Hospital Universitario La Paz, ALS Unit, Madrid
- Umeå University Hospital, Umeå, Sweden
- Leonard Wolfson Experimental Neurology Centre, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Arimoclomol (Open-label): 248 mg arimoclomol base 3 times daily (planned duration 152 weeks; actual duration after early termination of the trial approx. 28 weeks [range 2-71 weeks]).
Period: Overall Study
Arm/Group | Arimoclomol (Open-label)
Started | 120
Completed | 0
Not Completed | 120
Not completed — Adverse Event | 3
Not completed — Death | 22
Not completed — Withdrawal by Subject | 8
Not completed — Study terminated by sponsor | 87

BASELINE CHARACTERISTICS:
Groups:
- Arimoclomol (Open-label): 248 mg arimoclomol base 3 times daily
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 80
  More than one race | 0
  Unknown or Not Reported | 39
Region of Enrollment [Number; unit: participants]
  Canada | 2
  Netherlands | 10
  Sweden | 5
  Belgium | 5
  United States | 28
  Poland | 15
  Italy | 14
  United Kingdom | 2
  France | 17
  Germany | 7
  Spain | 15
ALS Functional Rating Scale - Revised (ALSFRS-R) [Mean (Standard Deviation); unit: units on a scale] — The ALSFRS-R is an ordinal rating scale used to determine subjects' subjective assessment of their capability and independence with 12 functional activities ('speech', 'salivation', 'swallowing', handwriting', 'cutting food and handling utensils', 'dressing and hygiene', 'turning in bed and adjusting bed clothes', 'walking', 'dyspnoea', 'orthopnoea' and 'respiratory insufficiency'). Each activity is rated on a 5-point scale (from 0 [no ability] to 4 [normal]), giving a maximal ALSFRS-R score of 48. A lower score corresponds to a lower capability and independence.
  units on a scale | 26.0 (10.38)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Over the Open-label Treatment Period
Description: Adverse event (AE) data were collected throughout the trial until early termination. The average duration of exposure was 198.7 days (approximately 28 weeks; standard deviation 99.57 days; minimum 16 days, maximum 494 days). 58 participants (48.3%) were exposed less than 6 months; 55 participants (45.8%) were exposed 6 to less than 12 months; 7 participants (5.8%) were exposed 12 to less than 18 months. No participant was treated for 76 weeks.
  Participants with on-treatment TEAEs are reported. An on-treatment TEAE is any TEAE in the on-treatment period defined as the time from first dose of IMP until 14 days since the last preceding administration of IMP (either before a temporary IMP interruption with duration >14 days or the last dose at the end of trial). A participant may have several on-treatment periods separated by interruption intervals.
Time Frame: From Day 1 in ORARIALS-02 to Early Termination, an average of approximately 28 weeks
Population: Safety analysis set: All enrolled patients who received at least one dose of arimoclomol.
Measure: Count of Participants; unit: Participants
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 120
Participants
  Treatment-emergent adverse events (TEAEs) | 93
  Mild TEAEs | 34
  Moderate TEAEs | 44
  Severe TEAEs | 15
  Treatment-related TEAEs | 31
  Probably related TEAEs | 9
  Possibly related TEAEs | 22
  Not related TEAEs | 62
  Serious TEAEs (SAEs) | 21
  Treatment-related serious TEAEs | 1
  TEAEs leading to IMP withdrawal | 9
  TEAEs leading to IMP interruption | 12

2. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Hematology (1)
Description: Standard hematology parameters. White blood cell differential count for basophils, eosinophils, leukocytes, lymphocytes, monocytes, and neutrophils, and platelet count.
Time Frame: Week 76
Population: Data only available for 2 participants at Week 76 since the trial was terminated early by the sponsor as a consequence of the results of ORARIALS-01 which did not meet any of its efficacy endpoints.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 2
10^9 cells/L
  Basophils, Week 76 | 0.030 (0.0000)
  Basophils, change from baseline to Week 76 | -0.015 (0.0071)
  Eosinophils, Week 76 | 0.150 (0.0141)
  Eosinophils, change from baseline to Week 76 | -0.070 (0.0424)
  Leukocytes, Week 76 | 9.120 (3.1537)
  Leukocytes, change from baseline to Week 76 | -0.565 (2.4395)
  Lymphocytes, Week 76 | 1.445 (0.4738)
  Lymphocytes, change from baseline to Week 76 | -0.365 (0.3041)
  Monocytes, Week 76 | 0.460 (0.1414)
  Monocytes, change from baseline to Week 76 | -0.055 (0.0212)
  Neutrophils, Segmented, Week 76 | 7.030 (3.4648)
  Neutrophils, Segmented, change from baseline to Week 76 | -0.070 (2.8001)
  Platelets, Week 76 | 334.0 (114.55)
  Platelets, change from baseline to Week 76 | 62.5 (103.94)

3. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Hematology (2)
Description: Standard hematology parameters. Percentage of leukocytes were determined for basophils, eosinophils, lymphocytes, monocytes, and neutrophils
Time Frame: Week 76
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of leukocytes
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 2
percentage of leukocytes
  Basophils/Leukocytes, Week 76 | 0.40 (0.141)
  Basophils/Leukocytes, change from baseline to Week 76 | -0.05 (0.212)
  Eosinophils/Leukocytes, Week 76 | 1.70 (0.424)
  Eosinophils/Leukocytes, change from baseline to Week 76 | -0.50 (0.849)
  Lymphocytes/Leukocytes, Week 76 | 17.85 (11.384)
  Lymphocytes/Leukocytes, change from baseline to Week 76 | -0.95 (8.132)
  Monocytes/Leukocytes, Week 76 | 5.05 (0.212)
  Monocytes/Leukocytes, change from baseline to Week 76 | -0.20 (1.556)
  Neutrophils/Leukocytes, Week 76 | 74.95 (12.092)
  Neutrophils/Leukocytes, change from baseline to Week 76 | 1.70 (10.607)

4. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Erythrocytes
Description: Standard hematology parameter.
Time Frame: Week 76
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 2
10^12 cells/L
  Erythrocytes, Week 76 | 3.70 (0.000)
  Erythrocytes, change from baseline to Week 76 | -0.40 (0.707)

5. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Hematocrit
Description: Standard hematology parameter.
Time Frame: Week 76
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L of cells / L of blood
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 2
L of cells / L of blood
  Hematocrit, Week 76 | 0.345 (0.0071)
  Hematocrit, change from baseline to Week 76 | -0.025 (0.0636)

6. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Hemoglobin
Description: Standard hematology parameter.
Time Frame: Week 76
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 2
g/L
  Hemoglobin, Week 76 | 115.5 (3.54)
  Hemoglobin, change from baseline to Week 76 | -14.0 (21.21)

7. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Clinical Chemistry (1)
Description: Standard clinical chemistry parameters. Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Creatine Kinase, Gamma Glutamyl Transferase, and Lactate Dehydrogenase.
Time Frame: Week 76
Population: Data only available for 1 participant at Week 76 since the trial was terminated early by the sponsor as a consequence of the results of ORARIALS-01 which did not meet any of its efficacy endpoints
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 1
U/L
  Alanine Aminotransferase, Week 76 | 14.0 (NA) — Standard deviation not applicable as N=1
  Alanine Aminotransferase, change from baseline to Week 76 | -31.0 (NA) — Standard deviation not applicable as N=1
  Alkaline Phosphatase, Week 76 | 97.0 (NA) — Standard deviation not applicable as N=1
  Alkaline Phosphatase, change from baseline to Week 76 | 16.0 (NA) — Standard deviation not applicable as N=1
  Aspartate Aminotransferase, Week 76 | 11.0 (NA) — Standard deviation not applicable as N=1
  Aspartate Aminotransferase, change from baseline to Week 76 | -15.0 (NA) — Standard deviation not applicable as N=1
  Creatine Kinase, Week 76 | 39.0 (NA) — Standard deviation not applicable as N=1
  Creatine Kinase, change from baseline to Week 76 | -118.0 (NA) — Standard deviation not applicable as N=1
  Gamma Glutamyl Transferase, Week 76 | 13.0 (NA) — Standard deviation not applicable as N=1
  Gamma Glutamyl Transferase, change from baseline to Week 76 | -15.0 (NA) — Standard deviation not applicable as N=1
  Lactate Dehydrogenase, Week 76 | 151.0 (NA) — Standard deviation not applicable as N=1
  Lactate Dehydrogenase, change from baseline to Week 76 | -42.0 (NA) — Standard deviation not applicable as N=1

8. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Clinical Chemistry (2)
Description: Standard clinical chemistry parameters. Calcium, Calcium Corrected, Cholesterol, Glucose, HDL Cholesterol, LDL Cholesterol, Potassium, Sodium, Triglycerides, and Urea Nitrogen.
Time Frame: Week 76
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 1
mmol/L
  Calcium, Week 76 | 2.220 (NA) — Standard deviation not applicable as N=1
  Calcium, change from baseline to Week 76 | -0.350 (NA) — Standard deviation not applicable as N=1
  Calcium Corrected, Week 76 | 2.270 (NA) — Standard deviation not applicable as N=1
  Calcium Corrected, change from baseline to Week 76 | -0.080 (NA) — Standard deviation not applicable as N=1
  Cholesterol, Week 76 | 3.050 (NA) — Standard deviation not applicable as N=1
  Cholesterol, change from baseline to Week 76 | -1.060 (NA) — Standard deviation not applicable as N=1
  Glucose, Week 76 | 8.50 (NA) — Standard deviation not applicable as N=1
  Glucose, change from baseline to Week 76 | 1.60 (NA) — Standard deviation not applicable as N=1
  HDL Cholesterol, Week 76 | 0.830 (NA) — Standard deviation not applicable as N=1
  HDL Cholesterol, change from baseline to Week 76 | -0.770 (NA) — Standard deviation not applicable as N=1
  LDL Cholesterol, Week 76 | 1.760 (NA) — Standard deviation not applicable as N=1
  LDL Cholesterol, change from baseline to Week 76 | -0.540 (NA) — Standard deviation not applicable as N=1
  Potassium, Week 76 | 3.90 (NA) — Standard deviation not applicable as N=1
  Potassium, change from baseline to Week 76 | -0.50 (NA) — Standard deviation not applicable as N=1
  Sodium, Week 76 | 138.0 (NA) — Standard deviation not applicable as N=1
  Sodium, change from baseline to Week 76 | -6.0 (NA) — Standard deviation not applicable as N=1
  Triglycerides, Week 76 | 1.100 (NA) — Standard deviation not applicable as N=1
  Triglycerides, change from baseline to Week 76 | 0.320 (NA) — Standard deviation not applicable as N=1
  Urea Nitrogen, Week 76 | 4.60 (NA) — Standard deviation not applicable as N=1
  Urea Nitrogen, change from baseline to Week 76 | -0.40 (NA) — Standard deviation not applicable as N=1

9. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Clinical Chemistry (3)
Description: Standard clinical chemistry parameters. Bilirubin, Creatinine, Direct Bilirubin, and Indirect Bilirubin.
Time Frame: Week 76
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 1
micromol/L
  Bilirubin, Week 76 | 5.0 (NA) — Standard deviation not applicable as N=1
  Bilirubin, change from baseline to Week 76 | -7.0 (NA) — Standard deviation not applicable as N=1
  Creatinine, Week 76 | 18.0 (NA) — Standard deviation not applicable as N=1
  Creatinine, change from baseline to Week 76 | -35.0 (NA) — Standard deviation not applicable as N=1
  Direct Bilirubin, Week 76 | 2.0 (NA) — Standard deviation not applicable as N=1
  Direct Bilirubin, change from baseline to Week 76 | -1.0 (NA) — Standard deviation not applicable as N=1
  Indirect Bilirubin, Week 76 | 3.0 (NA) — Standard deviation not applicable as N=1
  Indirect Bilirubin, change from baseline to Week 76 | -6.0 (NA) — Standard deviation not applicable as N=1

10. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Albumin and Protein
Description: Standard clinical chemistry parameters.
Time Frame: Week 76
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 1
g/L
  Albumin, Week 76 | 38.0 (NA) — Standard deviation not applicable as N=1
  Albumin, change from baseline to Week 76 | -13.0 (NA) — Standard deviation not applicable as N=1
  Protein, Week 76 | 64.0 (NA) — Standard deviation not applicable as N=1
  Protein, change from baseline to Week 76 | -16.0 (NA) — Standard deviation not applicable as N=1

11. Primary Outcome: Mean and Change From Baseline in Clinical Safety Laboratory Tests - Cystatin C
Description: Standard clinical chemistry parameter.
Time Frame: Week 76
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 2
mg/L
  Cystatin C, Week 76 | 1.310 (0.7495)
  Cystatin C, change from baseline to Week 76 | 0.350 (0.6364)

12. Primary Outcome: Mean and Change From Baseline in Vital Signs - Blood Pressure
Description: Standard vital signs. Systolic and diastolic blood pressure.
Time Frame: Week 76
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 1
mmHg
  Systolic Blood Pressure, Week 76 | 112.0 (NA) — Standard deviation not applicable as N=1
  Systolic Blood Pressure, change from baseline to Week 76 | -10.0 (NA) — Standard deviation not applicable as N=1
  Diastolic Blood Pressure, Week 76 | 76.0 (NA) — Standard deviation not applicable as N=1
  Diastolic Blood Pressure, change from baseline to Week 76 | -1.0 (NA) — Standard deviation not applicable as N=1

13. Primary Outcome: Mean and Change From Baseline in Vital Signs - Pulse Rate
Description: Standard vital signs measurement.
Time Frame: Week 76
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 1
beats/min
  Pulse Rate, Week 76 | 86.0 (NA) — Standard deviation not applicable as N=1
  Pulse Rate, change from baseline to Week 76 | -3.0 (NA) — Standard deviation not applicable as N=1

14. Primary Outcome: Mean and Change From Baseline in Vital Signs - Respiratory Rate
Description: Standard vital signs measurement.
Time Frame: Week 76
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 1
breaths/min
  Respiratory Rate, Week 76 | 12.0 (NA) — Standard deviation not applicable as N=1
  Respiratory Rate, change from baseline to Week 76 | -4.0 (NA) — Standard deviation not applicable as N=1

15. Primary Outcome: Mean and Change From Baseline in Vital Signs - Temperature
Description: Standard vital signs measurement.
Time Frame: Week 76
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 1
Degrees Celsius
  Temperature, Week 76 | 36.40 (NA) — Standard deviation not applicable as N=1
  Temperature, change from baseline to Week 76 | 0.80 (NA) — Standard deviation not applicable as N=1

16. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities in Clinical Safety Laboratory Tests and Vital Signs Over the Open-label Treatment Period
Description: Clinical safety laboratory data and vital signs were collected throughout the trial until early termination. The average duration of exposure was 198.7 days (approximately 28 weeks; standard deviation 99.57 days; minimum 16 days, maximum 494 days). 58 participants (48.3%) were exposed less than 6 months; 55 participants (45.8%) were exposed 6 to less than 12 months; 7 participants (5.8%) were exposed 12 to less than 18 months. No patient was treated for 76 weeks.
Time Frame: From Day 1 in ORARIALS-02 to Early Termination, an average of approximately 28 weeks
Population: Safety analysis set: All enrolled patients that received at least one dose of arimoclomol.
Measure: Count of Participants; unit: Participants
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 120
Participants
  Hemoglobin (g/L) <= 95 (Females) <= 115 (Males) | 10
  Hemoglobin (g/L) >= 165 (Females), >= 185 (Males) | 0
  Erythrocytes (10^12/L) <= 3.5 (Females), <= 3.8 (Males) | 16
  Erythrocytes (10^12/L) >= 6.0 (Females), >= 7.0 (Males) | 0
  Hematocrit <= 0.32 (Females), <= 0.37 (Males) | 21
  Hematocrit >= 0.5 (Females), >= 0.55 (Males) | 0
  Leukocytes (10^9/L) <= 2.8 | 0
  Leukocytes (10^9/L) >= 16 | 3
  Neutrophils/Leukocytes (%) <= 20 | 0
  Neutrophils/Leukocytes (%) >= 85 | 3
  Eosinophils/Leukocytes (%) >= 10 | 1
  Basophils/Leukocytes (%) >= 10 | 0
  Lymphocytes/Leukocytes (%) <= 10 | 6
  Lymphocytes/Leukocytes (%) >= 75 | 0
  Monocytes/Leukocytes (%) >= 15 | 0
  Platelets (10^9/L) <= 75 | 0
  Platelets (10^9/L) >= 600 | 0
  Aspartate Aminotransferase (U/L) >= 3 x Upper Limit of Normal (ULN) | 0
  Alanine Aminotransferase (U/L) >= 3 x ULN | 7
  Bilirubin (umol/L) >= 34 | 2
  Direct Bilirubin (umol/L) >= 12 | 0
  Indirect Bilirubin (umol/L) >= 22 | 4
  Alkaline Phosphatase (U/L) >= 3 x ULN | 1
  Gamma Glutamyl Transferase (U/L) >= 200 | 4
  Creatinine (umol/L) >= 1.5 x ULN | 1
  Urea Nitrogen (mmol/L) >= 11 | 7
  Sodium (mmol/L) <= 125 | 2
  Sodium (mmol/L) >= 155 | 1
  Potassium (mmol/L) <= 3.0 | 4
  Potassium (mmol/L) >= 6.0 | 0
  Calcium (mmol/L) <= 1.8 | 0
  Calcium (mmol/L) >= 3.0 | 2
  Glucose (mmol/L) <= 3.9 (Fasting=No or blank) | 8
  Glucose (mmol/L) >= 11.1 (Fasting=No or blank) | 7
  Glucose (mmol/L) <= 3.5 (Fasting=Yes) | 0
  Glucose (mmol/L) >= 7.0 (Fasting=Yes) | 7
  Protein (g/L) <= 45 | 1
  Protein (g/L) >= 95 | 0
  Albumin (g/L) <= 27 | 2
  Cholesterol (mmol/L) >= 7.8 (Fasting=No or blank) | 15
  Cholesterol (mmol/L) >= 6.2 (Fasting=Yes) | 15
  Triglycerides (mmol/L) >= 5.65 (Fasting=No or blank) | 6
  Triglycerides (mmol/L) >= 4.2 (Fasting=Yes) | 3
  LDL Cholesterol (mmol/L) >= 5.3 (Fasting=No or blank) | 13
  LDL Cholesterol (mmol/L) >= 4.9 (Fasting=Yes) | 7
  HDL Cholesterol (mmol/L) <= 0.8 (Fasting=No or blank) | 11
  HDL Cholesterol (mmol/L) <= 0.9 (Fasting=Yes) | 2
  Creatine Kinase (U/L) >= 400 (Females) >= 750 (Males) | 20
  Lactate Dehydrogenase (U/L) >= 750 | 0
  Pulse Rate <50 and decrease from baseline of >= 15 beats/min | 0
  Pulse Rate >120 and increase from baseline of >= 15 beats/min | 0
  Diastolic Blood Pressure <=50 and decrease from baseline of >= 15 mmHg | 1
  Diastolic Blood Pressure >105 and increase from baseline of >= 15 mmHg | 6
  Systolic Blood Pressure <=90 and decrease from baseline of >= 20 mmHg | 3
  Systolic Blood Pressure >180 and increase from baseline of >= 20 mmHg | 0

17. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS) Over the Open-label Treatment Period
Description: The C-SSRS is a detailed questionnaire assessing both suicidal behavior and suicidal ideation through a series of simple, plain-language questions administered as an interview by a qualified investigator or delegate.
Time Frame: From Day 1 in ORARIALS-02 to Early Termination, an average of approximately 28 weeks
Population: Safety analysis set: All enrolled patients who received at least one dose of arimoclomol.
Measure: Count of Participants; unit: Participants
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 120
Participants
  Suicidal ideation (yes on any 1 of the following 5 items) | 16
  Wish to be Dead | 15
  Non-specific active suicidal thoughts | 10
  Active Suicidal ideation with any methods (not Plan) without intent to Act | 5
  Active suicidal ideation with some intent, without Specific Plan | 1
  Active Suicidal ideation with specific Plan and Intent | 0
  Suicidal Behavior (yes on any 1 of the following 5 items) | 0
  Preparatory acts or behavior | 0
  Aborted Attempt | 0
  Interrupted Attempt | 0
  Actual Attempt (non-fatal) | 0
  Completed Suicide | 0
  Suicidal ideation or Behavior (yes to any of the above 10 items) | 16
  Self-injurious Behavior without suicidal intent | 0

18. Secondary Outcome: Change in ALS Functional Rating Scale - Revised (ALSFRS-R) From Baseline to Week 76
Description: The ALSFRS-R is an ordinal rating scale used to determine subjects' subjective assessment of their capability and independence with 12 functional activities ('speech', 'salivation', 'swallowing', handwriting', 'cutting food and handling utensils', 'dressing and hygiene', 'turning in bed and adjusting bed clothes', 'walking', 'dyspnoea', 'orthopnoea' and 'respiratory insufficiency'). Each activity is rated on a 5-point scale (from 0 [no ability] to 4 [normal]), giving a maximal ALSFRS-R score of 48. A lower score corresponds to a lower capability and independence.
Time Frame: Week 76
Population: Data were not collected at Week 76 since the trial was terminated early by the sponsor as a consequence of the results of ORARIALS-01 which did not meet any of its efficacy endpoints.
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 0

19. Secondary Outcome: Change in Percentage (%) Predicted Slow Vital Capacity (SVC) From Baseline to Week 76 (for Subjects Who Did Not Meet the Survival Endpoint in the ORARIALS-01 Trial)
Description: Slow vital capacity (SVC) measures the volume that can be exhaled from a full inhalation after exhaling to a maximum as slowly as possible. Predicted SVC was derived per European Community of Coal and Steel (ECCS) reference equations:
  * If male: Predicted SVC = 0.061 x height (cm) - 0.028 x age (years) - 4.65
  * If female: Predicted SVC = 0.0466 x height (cm) - 0.024 x age (years) - 3.28
Time Frame: 76 weeks
Population: Data only available for 1 patient at Week 76 since the trial was terminated early by the sponsor as a consequence of the results of ORARIALS-01 which did not meet any of its efficacy endpoints.
Measure: Mean (Standard Deviation); unit: percentage of predicted SVC
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 1
percentage of predicted SVC | -21.6 (NA) — Standard deviation not applicable as N=1

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected throughout the trial until early termination. The average duration of exposure was 198.7 days (approximately 28 weeks; standard deviation 99.57 days; minimum 16 days, maximum 494 days). 58 participants (48.3%) were exposed less than 6 months; 55 participants (45.8%) were exposed 6 to less than 12 months; 7 participants (5.8%) were exposed 12 to less than 18 months.
Description: A treatment-emergent AE (TEAE) is defined as an AE with onset, or a pre-existing AE that worsened in severity, on or after the first dose of IMP. An on-treatment TEAE is any TEAE in the on-treatment period defined as the time from first dose of IMP until 14 days since the last preceding administration of IMP (either before a temporary IMP interruption with duration >14 days or the last dose at the end of trial). A patient may have several on-treatment periods separated by interruption intervals.
Arm/Group | Arimoclomol (Open-label)
All-Cause Mortality (participants affected / at risk) | 23/120
Serious Adverse Events (participants affected / at risk) | 21/120
Other Adverse Events (participants affected / at risk) | 91/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arimoclomol (Open-label) (N=120)
Pneumonia (Infections and infestations) | 7
Clostridium difficile infection (Infections and infestations) | 1
Corona virus infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
False positive investigation result (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arimoclomol (Open-label) (N=120)
Urinary tract infection (Infections and infestations) | 7
Corona virus infection (Infections and infestations) | 6
Constipation (Gastrointestinal disorders) | 8
Fall (Injury, poisoning and procedural complications) | 8
Cystatin C increased (Investigations) | 7
Anaemia (Blood and lymphatic system disorders) | 6
Fungal skin infection (Infections and infestations) | 3
Flatulence (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 5
Head injury (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 3
Tachycardia (Cardiac disorders) | 3
Hypertension (Vascular disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3

LIMITATIONS AND CAVEATS:
Early termination led to data for a limited number of patients. No conclusions can be drawn from the laboratory results due to data for only a few patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03836716/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03836716/SAP_001.pdf